CLINICAL TRIAL: NCT06685302
Title: Effect of Adding Ultrasound-guided Percutaneous Neuromodulation to Conventional Treatment of Ultrasound-guided Percutaneous Electrolysis and Eccentric Exercises in Patients With Patellar Tendinopathy. Randomized Clinical Trial
Brief Title: Addition of Ultrasound-guided Percutaneous Neuromodulation to Ultrasound-guided Percutaneous Electrolysis and Eccentric Exercises in Patellar Tendinopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Dr. Pablo Herrero Gallego, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNM, PES and EE in PT. ECA
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Patellar Tendinitis; Patella; Tendinitis; Patellar Tendinopathy / Jumpers Knee
Keywords: percutaneous neuromodulation; percutaneous electrolysis; eccentric exercise; patellar tendinopathy; jumper´s knee
MeSH Terms: conditions — Patella Fracture; Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-PNM + US-PE + EE (Experimental): Patients receive three interventions: ultrasound-guided percutaneous neuromodulation, ultrasound-guided percutaneous electrolysis and eccentric exercises
  Interventions: Other: US-guided PNM; Other: US-guided PE
- US-PE + EE (Active Comparator): Patients receive two interventions: ultrasound-guided percutaneous electrolysis and eccentric exercises
  Interventions: Other: US-guided PE; Other: EE

INTERVENTIONS:
Other: US-guided PNM — The patient will be positioned in supine with approximately 20 degrees of knee flexion, supported by a cushion. The treatment area is sterilized in advance with 2% chlorhexidine, and new needles and ultrasound probe covers are used for each intervention. The femoral nerve is targeted under ultrasound guidance, just distal to the inguinal ligament, with an electrode patch placed on the patellar tendon to complete the circuit. A current of 2 Hz, 250 μs pulse width, and variable intensity is applied to reach the patient's comfortable contraction threshold without inducing pain, for a duration of 25 minutes, following the protocol established by MVClinic Institute. This intervention will be performed on the first day, at 7 days, and at 14 days, following the previously mentioned protocol.
  Arms: US-PNM + US-PE + EE
Other: US-guided PE — The patient will be positioned in supine with approximately 20º of knee flexion, supported by a cushion. Prior to the EP procedure, the treatment area will be sterilized with 2% chlorhexidine, and new needles and ultrasound probe covers will be used for each session. Three EP interventions will be performed under ultrasound guidance following the protocol developed by MVClinic Institute (2) for treating tendinopathies, using a longitudinal, long-axis view of the patellar tendon. A galvanic current of 3 mA will be applied for 3 seconds, with slight three-dimensional adjustments in needle placement after each impact to administer a total of 3 impacts on the target tissue. This intervention will be performed on the first day, at 7 days, and at 14 days, following the previously mentioned protocol.
Other: EE — Three sets of 15 repetitions of single-leg squats on a 25º inclined plane, performed twice daily, following Young's protocol for patellar tendinopathies. The speed of execution may be increased as long as, if there is pain during the exercise, it does not exceed a 2-3 on the VAS scale.
  Arms: US-PE + EE

SUMMARY:
Patellar tendinopathy, or "jumper's knee," is a prevalent condition involving patellar tendon degeneration due to structural overuse, common among athletes, particularly males over 18 in sports like volleyball, basketball, or football. It causes tendon thickening, collagen disorganization, fibroblast proliferation, neovascularization, and neurogenesis. Symptoms include anterior knee pain that worsens with activity, tenderness at the proximal tendon insertion, and functional limitations. Diagnosis often utilizes ultrasound imaging. While surgical treatment is reserved for severe cases, non-surgical options prioritize physiotherapy-especially eccentric exercises and newer invasive techniques like percutaneous electrolysis and neuromodulation. However, there is still no research on the effects when combining these three treatment options.

DETAILED DESCRIPTION:
Patellar tendinopathy, also known as "jumper's knee," is one of the most common conditions affecting the patellar tendon. It involves degeneration of the tendon, primarily due to excessive structural overuse. This condition leads to various changes within the tissue, including tendon thickening, collagen fiber degeneration and disorganization, disruption in the parallel alignment of healthy collagen fibers, fibroblast proliferation with incomplete injury repair, neovascularization, and neurogenesis. Various studies indicate a high prevalence of patellar tendinopathy among athletes and the general population, with rates of 0.1% and 18.3%, respectively. The condition is more frequently observed in males over 18 who participate in sports such as volleyball, basketball, or football.

Clinical symptoms of patellar tendinopathy include anterior knee pain that worsens with exercise, post-exercise, or during prolonged knee flexion; localized pain and tenderness at the proximal tendon insertion; and functional impairment in actions such as squatting with ankle plantar flexion.There are different diagnostic methods, both medical and physiotherapeutic, to determine the presence of patellar tendinopathy. In this context, imaging evaluations through ultrasound show potential as diagnostic and follow-up tool.

Only in advanced stages of tendon degeneration is surgical treatment considered, which may involve open surgery or arthroscopy. Among non-surgical treatments for patellar tendinopathy, medical options focus on platelet-rich plasma injections, hyaluronic acid, nonsteroidal anti-inflammatory drugs, or corticosteroids. However, conservative physiotherapy is typically the first choice, generally based on eccentric exercises, and invasive techniques such as percutaneous electrolysis or percutaneous neuromodulation.

Current literature provides evidence supporting percutaneous electrolysis, percutaneous neuromodulation and eccentric exercises as therapeutic methods for tendinopathies. However, there is presently no evidence or studies regarding the combination of these three techniques.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 50 years
* Experiencing localized anterior knee pain at the lower pole of the patella for at least two weeks
* Engaging in any type of sport at least three times per week
* Scoring less than 80 points on the VISA-P questionnaire in its Spanish version
* Having carefully read and signed the study's informed consent form

Exclusion Criteria:

* Any contraindication for invasive techniques (such as belonephobia, allergies to materials used, cancer, thrombophlebitis, skin conditions, or febrile states)
* Any lower limb pathology or severe chronic condition (e.g., Osgood-Schlatter syndrome or Sinding-Larsen-Johansson syndrome)
* Pharmacological treatment within the 48 hours prior to the intervention
* Knee surgeries within the past year
* Corticosteroid injections within the previous 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Pain | Measurements will be conducted on day 1, 7, 14, 21 and 28
  This will be measured using the Visual Analog Scale (VAS). Minimum and maximum values are 1-10, being 10 worst possible pain

SECONDARY OUTCOMES:
Pain and Functionality | Measurements will be conducted on days 1 and 28
  This will be measured using the VISA-P questionnaire
Quality of Life | Measurements will be conducted on days 1 and 28
  This will be measured using the SF-36 questionnaire
Functionality | Measurements will be conducted on days 1 and 28
  This will be measured using the pistol squat exercise
Tendinous tissue condition | Measurements will be conducted on days 1 and 28
  This will be measured using ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero, Physiotherapist, Study Director — Universidad de Zaragoza
Locations (1):
- University of Zaragoza, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a reasonable request contacting with the main author once data has been published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once research has been published
Access Criteria: Study protocol will be publish in a scientific journal